CLINICAL TRIAL: NCT02088788
Title: Reduction in Physician Radiation Exposure During Radial Access Cardiac Catheterization Using a Radiation Protection Board
Brief Title: Physician Radiation Exposure During Radial Access Cardiac Catheterization Using a RAD Board
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, James C. Blankenship, Director of Cardiology, Geisinger Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2013-0140
Record Dates: First submitted 2014-03-13; First posted 2014-03-17 (Estimated); Results first posted 2018-10-24 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-09

CONDITIONS: Radiation Exposure to Operator
Keywords: radiation; radiation injury; occupational risk
MeSH Terms: conditions — Radiation Injuries | interventions — Communication Devices for People with Disabilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Board (Rad Board") (Experimental): Radial artery catheterization is performed using radio-opaque armboard
  Interventions: Device: Board
- No Board (Active Comparator): Regular radio-penetrating armboard is used (the one normally used during non-study procedures) with a radio-opaque pelvic shield
  Interventions: Device: No Board

INTERVENTIONS:
Device: Board — Also has radio-dense pelvic shielding
  Other Names: "Rad Board"
  Arms: Board (Rad Board")
Device: No Board — Radio-lucent armboard for radial access with radio-dense drape across pelvis
  Arms: No Board

SUMMARY:
Radiation exposure to operator is an occupational hazard of invasive cardiologists. During radial access for diagnostic catheterization, a new radio-dense arm board is advertised to reduce operator radiation exposure. The investigators randomize patients to a new radio-dense armboard versus a standard radio-transparent armboard during diagnostic catheterization and measure radiation exposure to the operator. Both groups have a radio-dense pelvic shield in place. The investigators hypothesize that operator radiation dose will be decreased by use of the radio-dense armboard.

DETAILED DESCRIPTION:
Hypothesis:

Compared to standard shielding with a lead pelvic drape alone, using a radio-opaque arm board in addition to the pelvic drape will decrease operator radiation exposure during radial access cardiac catheterization by at least 30%.

STUDY DESIGN This is a randomized, prospective study where patients will be randomized by random numbers in sealed envelopes to standard shielding (pelvic drape alone, the "no-board group") or to experimental shielding (pelvic drape plus radiation board, the "board group").

A robust radiation safety monitoring program is in place. Patient exposure is measured by the catheterization laboratory equipment and recorded. Lindauer Microstar Nanodot badges worn at waist level above the radiation lead will be used to measure operator radiation exposure. A new Nanodot will be used for every case. Radiation exposure to the operator's Nanodot will be measured immediately after each procedure by a technician blinded to study assignment.

All patients 18-89 years old presenting to Geisinger Medical Center for diagnostic cardiac catheterization will be evaluated for the study. All interventional or diagnostic cardiologists and fellows that will be performing the cardiac catheterization procedure also will be study subjects. Approximately 215 Geisinger patients who satisfy inclusion and exclusion criteria will be included. Approximately 6 interventional cardiologists, 2 diagnostic cardiologists and 10 fellows will be included in this study.

ELIGIBILITY:
Inclusion Criteria:

Operators: Interventional or diagnostic interventional attendings and fellows, operators willing to participate.

Patients: Age 18-89 years old requiring catheterization at Geisinger Medical Center using radial access

Exclusion Criteria:

* patients with CABG, requiring extensive imaging, with operator switch during the procedure
* patients in whom the procedure took unusual time because of anatomic issues, and need to switch to alternative access.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2013-06; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James C Blankenship, MD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Medical Center, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Board (Rad Board") | No Board
Started | 135 | 130
Completed | 105 | 89
Not Completed | 30 | 41

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Board (Rad Board") | No Board | Total
Number analyzed (Participants) | 105 | 89 | 194
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (12.1) | 64.2 (9.5) | 64.5 (10.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 38 | 75
  Male | 68 | 51 | 119
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Operator Radiation Exposure
Description: mSieverts radiation dose to the operator during diagnostic catheterization
Time Frame: during initial diagnostic catheterization procedure, an average of 30 minutes
Measure: Median (Inter-Quartile Range); unit: mSv
Arm/Group | Board (Rad Board") | No Board
Number analyzed (Participants) | 105 | 89
mSv | .65 [.57 to .78] | .56 [.48 to .63]

2. Secondary Outcome: Radiation Exposure to Operator During Diagnostic Catheterization With Versus Without Ventriculography/Aortography
Description: mSieverts radiation dose to the operator during diagnostic catheterization with versus without ventriculography/aortography. This outcome measure includes 2 types of procedures: diagnostic catheterization plus LV gram and diagnostic catheterization plus aortography. Ventriculography is defined as injection through a pigtail catheter into the left ventricle using a power injector. Aortography is defined as injection through a pigtail catheter into the aorta using a power injector.
Time Frame: During procedure, an average of 35 minutes
Measure: Median (Inter-Quartile Range); unit: mSv
Arm/Group | Board (Rad Board") | No Board
Number analyzed (Participants) | 105 | 89
mSv
  With Ventriculogram/aortogram | .65 [.55 to .78] | .61 [.5 to .66]
  Without ventriculogram/aortogram | .66 [.58 to .79] | .54 [.48 to .61]

ADVERSE EVENTS:
Time Frame: Adverse events were not collected for this study. Consent was not obtained from patients since no experimental procedures involved patients.
Description: Adverse events were not collected for this study.
Arm/Group | Board (Rad Board") | No Board
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
We excluded post hoc procedures that required prolonged imaging. This resulted in unequal sizes of the board and no-board groups. As a single-center trial, results may not be generalizable to cath labs with different radiation protection set-ups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes